CLINICAL TRIAL: NCT04229095
Title: Medication Development for Protracted Abstinence in Alcoholism: Suvorexant Versus Placebo
Brief Title: Medication Development in Alcoholism: Suvorexant Versus Placebo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Scripps Research Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: P60AA006420 (NIH); P60AA006420 (NIH)
Record Dates: First submitted 2020-01-09; First posted 2020-01-14 (Actual); Results first posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Alcohol Use Disorder (AUD)
MeSH Terms: conditions — Alcoholism | interventions — suvorexant; Sugars

STUDY DESIGN:
Intervention Model Description: Parallel Assignment, Double-Blind, Randomized Stratified at randomization based on sex and Pittsburgh Sleep Quality Index Total Score (PSQI) greater than or equal to 5 versus less than 5.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Belsomra,(suvorexant) (Active Comparator): 20 mg single-dose administration given on an inpatient clinical research unit
  Interventions: Drug: Suvorexant 20 mg
- Placebo (Placebo Comparator): Placebo single-dose administration given on an inpatient clinical research unit
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Suvorexant 20 mg — Single-dose administration of 20 mg suvorexant given on an inpatient clinical research unit
  Other Names: Belsomra
  Arms: Belsomra,(suvorexant)
Drug: Placebo oral tablet — Single-dose administration of placebo given on an inpatient clinical research unit
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The primary hypotheses under test are that alcohol dependent subjects treated with suvorexant will report decreased craving for alcohol following alcohol exposure in the laboratory and report significantly less drinking under naturalistic conditions, than those treated with placebo. Suvorexant (Belsomra®) received approval by the FDA in 2014 for treatment of insomnia. To control for any effect of pre-existing sleep disturbance for which suvorexant may be indicated, subjects will be stratified on the basis of a Pittsburgh Sleep Quality Index total score of > 5 versus <5. Subjects were also stratified by sex.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers, 18-65 years of age.
* Meets Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for current alcohol use disorder of moderate or greater severity (AUD-MS).
* In the month prior to screening, reports drinking ≥ 21 standard drinks per week if male, ≥ 14 if female, with at least one heavy drinking day (≥ 5 males, ≥ 4 females) per week.
* Subjects will not be seeking treatment because the medication studies are not treatment trials, and to avoid exposing treatment-seekers to alcohol cues
* Subjects must be abstinent a minimum of 3 days (but not more than 7 days) prior to the human lab session.
* Negative blood alcohol content (BAC) and a Clinical Institute Withdrawal Assessment (CIWA) score of < 9 at time of randomization and lab session to eliminate acute alcohol or withdrawal effects on dependent measures.
* In acceptable health in the judgment of the study physician, on the basis of interview, medical history, physical exam, EKG, routine urine and blood chemistry.
* Subjects with a history of depression, who have been on a stable dose of anti-depressant medication for at least 3 months, and do not meet current DSM-5 criteria for depression or anxiety.
* Females with childbearing potential must have a negative pregnancy test on the screening and randomization visits and agree to use effective birth control for the duration required by a given study.
* Able to provide informed consent and understand questionnaires and study procedures in English.
* Willing to comply with the provisions of the protocol and take oral medication.

Exclusion Criteria:

* Meets DSM-5 criteria for a major psychiatric disorder, including mood or anxiety disorders or substance use disorders other than alcohol or nicotine, or, mild cannabis use disorder
* Has a urine drug screen (UDS) positive for substances of abuse other than alcohol or marijuana
* Significant medical disorders that will increase potential risk or interfere with study participation as determined by the study physician.
* Liver function tests more than 3 times the upper limit of normal or elevated bilirubin.
* Subjects taking digoxin or CYP3A inhibitors or inducers, metabolism by CYP3A is the major elimination pathway for suvorexant.
* Treatment within the month prior to screening with (1) an investigational drug, (2) medications which may negatively interact with study medications, or (3) drugs that may influence study outcomes (e.g., disulfiram [Antabuse], naltrexone [ReVia], acamprosate [Campral], or anticonvulsants).
* Ongoing treatment with medications that may increase risk, including prescribed, over-the-counter, and herbal preparations, as determined by the study physician.
* Sexually active female subjects with childbearing potential who are pregnant, nursing, or refuse to use effective methods of birth control for the duration of the study.
* No fixed domicile and/or no availability by home or mobile telephone.
* History of hypersensitivity to the study drug or the ingredients.
* Failure to take double-blind medication as prescribed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. Mason, Ph.D., Principal Investigator — The Scripps Research Institute
Locations (1):
- Scripps Research, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited for study participation at the Laboratory of Clinical Psychopharmacology at The Scripps Research Institute in La Jolla, California from 09/30/2021-11/08/2022.
Pre-assignment Details: Thirty-two subjects did not meet admission criteria and 12 subjects declined participation.
Groups:
- Placebo, (Sugar Pill): Placebo single-dose administration given on an inpatient clinical research unit
  Placebo oral tablet: Single-dose administration of placebo given on an inpatient clinical research unit
Period: Overall Study
Arm/Group | Belsomra,(Suvorexant) | Placebo, (Sugar Pill)
Started | 14 | 12
Completed | 14 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belsomra,(Suvorexant) | Placebo, (Sugar Pill) | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.29 (11.7) | 38.83 (11.0) | 37.46 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 6 | 9 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 8 | 17
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 12 | 26
DSM-V symptom Count [Mean (Standard Deviation); unit: symptom count] — Symptom count from the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) criteria for Alcohol Use Disorder (AUD)
  symptom count | 6.43 (2.1) | 8.08 (2.0) | 7.19 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS) of Craving Severity: 2 Arms
Description: VAS to alcohol cues minus VAS to water cues on a 0-20 VAS scale. Higher scores indicate greater craving strength with a minimum score of 0 and a maximum score of 20.
Time Frame: 1 hour during cue reactivity session
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Belsomra,(Suvorexant) | Placebo
Number analyzed (Participants) | 14 | 12
score on a scale | 2.38 (0.90) | 1.44 (0.62)

2. Primary Outcome: Visual Analog Scale (VAS) Strength of Craving: Combined Arms Conditional Model
Description: as for outcome 1
Time Frame: 1 hour during cue reactivity session
Population: All randomized subjects
Measure: Number; unit: score on a scale
Groups:
- Combined Drug/Placebo Condition: The drug and placebo groups were combined for the purposes of the mixed effect model analysis specified in the statistical analysis plan for the primary outcome analysis.
Arm/Group | Combined Drug/Placebo Condition
Number analyzed (Participants) | 26
score on a scale | .94
Statistical Analysis 1: Comparison: Combined Drug/Placebo Condition; Mixed effect model with directional hypothesis that drug reduces strength of craving (VAS). Principle predictors were drug condition, and baseline sleep disturbance (Pittsburgh Sleep Quality Index {PSQI} total score less than 5 or 5 and greater). Arms were combined for this analysis; Test type: Superiority; p = .007, Mixed Models Analysis; Slope = -4.58, 95% CI 1-sided [upper limit -1.01], Standard Error of Mean 1.82 — The effect of the drug on lowering VAS was limited to individuals with impaired sleep at baseline (PSQI > or = to 5)

3. Secondary Outcome: Number of Standard Drinks Per Day: 2 Arms
Description: Number of standard drinks per day using the Timeline Followback Interview (TLFB). Total number of alcohol drinks consumed per day with a minimum value of 0 and an undetermined maximum value
Time Frame: Up to one week following single dose administration
Measure: Mean (Standard Error); unit: Standard drinks per day
Arm/Group | Belsomra,(Suvorexant) | Placebo, (Sugar Pill)
Number analyzed (Participants) | 14 | 12
Standard drinks per day | 3.59 (0.87) | 3.46 (0.88)

4. Secondary Outcome: Number of Standard Drinks Per Day: Combined Arms Conditional Model
Description: Number of standard drinks per day using the Timeline Followback Interview (TLFB). Total number of alcoholic drinks consumed per day with a minimum value of 0 and an undetermined maximum value.
Time Frame: Up to one week following single dose administration
Population: Of the 26 subjects randomized, all 17 subjects that had any follow up drinking data were included in this analysis.
Measure: Number; unit: number of standard drinks per day
Arm/Group | Combined Drug/Placebo Condition
Number analyzed (Participants) | 17
number of standard drinks per day | -1.52
Statistical Analysis 1: Comparison: Combined Drug/Placebo Condition; Mixed effect model with directional hypothesis that drug reduces number of drinks per day. Principle predictors were drug condition and sex. Arms were combined for this analysis; Test type: Superiority; p = .0025, Mixed Models Analysis; Mean Difference (Net) = -1.52, 95% CI 1-sided [upper limit -0.46], Standard Error of Mean 0.54

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at all study visits, for any average duration of 3 weeks.
Description: Adverse events, both serious and other, were documented at all study visits by the Medical Assistant on the adverse event case report form.
Arm/Group | Belsomra,(Suvorexant) | Placebo, (Sugar Pill)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 8/14 | 7/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belsomra,(Suvorexant) (N=14) | Placebo, (Sugar Pill) (N=12)
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0
Feeling cold (General disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 1
Somnolence (Nervous system disorders) | 4 | 3
Vivid dreams (Nervous system disorders) | 1 | 0
Mental fatigue (Psychiatric disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
The actual enrollment was 26 subjects, relative to the planned enrollment of 50 subjects, due to chronic staffing problems for overnight studies at the Altman Clinical and Translational Research Institute (ACTRI) at the University of California-San Diego (UCSD) that resulted in multiple pre-randomization visit cancellations. Alternative inpatient beds were not available at general hospitals due to the prioritization of their facilities for COVID-19 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT04229095/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT04229095/SAP_001.pdf
  • Informed Consent Form (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT04229095/ICF_002.pdf